CLINICAL TRIAL: NCT00069992
Title: Safety And Efficacy of Sub-Myeloablative Allogeneic Stem Cell Transplantation For Patients With Myeloproliferative Disorder (MPD), Myelodysplastic Syndrome (MDS), Acute Myelogenous Leukemia (AML) or Chronic Myelogenous Leukemia
Brief Title: Total-Body Irradiation, Fludarabine, and Alemtuzumab Followed By Stem Cell Transplant in Treating Patients With Myeloproliferative Disorder, MS, AML, or CML
Acronym: MPDMDSBMT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Closed due to competing protocols
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other); Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, George Carrum, Associate Professor; Director-Adult Outpatient Clinic, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-10857-MPDMDSBMT
Record Dates: First submitted 2003-10-03; First posted 2003-10-07 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-10

CONDITIONS: Chronic Myeloproliferative Disorders; Leukemia; Myelodysplastic Syndromes
Keywords: polycythemia vera; essential thrombocythemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; primary myelofibrosis; chronic myelogenous leukemia; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); childhood myelodysplastic syndromes
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Myelodysplastic Syndromes; Polycythemia Vera; Thrombocythemia, Essential; Primary Myelofibrosis; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Congenital Abnormalities | interventions — Whole-Body Irradiation; fludarabine; fludarabine phosphate; Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Submyeloablative Allogeneic Stem Cell Transplant (Experimental): Total Body Irradiation Fludarabine Campath 1H
  Interventions: Radiation: Total Body Irradiation; Drug: Fludarabine; Drug: Campath 1H

INTERVENTIONS:
Radiation: Total Body Irradiation — Total body irradiation of 450cGy as a single dose, day -6
  Other Names: TBI
Drug: Fludarabine — Fludarabine 30mg/m2 Day -5 to -2
  Other Names: Fludara
Drug: Campath 1H — Campath 1H dosing as per institutional SOPs Day -5 to -2
  Other Names: Alemtuzumab

SUMMARY:
Patients are being asked to participate in this study because they have a malignant blood disease such as Myelodysplastic Syndrome (MDS), Myeloproliferative Disorder (MPD), Acute Myelogenous Leukemia (AML) or Chronic Myelogenous Leukemia (CML). We feel that patients could benefit from an allogeneic (meaning the cells come from a donor other than themself) stem cell transplant. The donor would be a family member or an unrelated person that is felt to be a good match for the patient. Stem cells are cells that are made in the bone marrow (spongy material that fills the middle of the bones). As the stem cells grow, they change into different types of blood cells that they need. This includes red blood cells that carry oxygen around the body, white blood cells that help to fight infections, and platelets that help to prevent and stop bleeding. Usually, patients are given high doses of chemotherapy before a stem cell transplant. High doses of chemo destroy the bone marrow. Healthy stem cells from a donor are then given to replace the patient's unhealthy cells. However, because of complications with the patient's disease, they have a high risk of having life-threatening side effects. These include serious damage to organs such as the lung, liver, kidney and heart. There is also an increased risk of bacterial, fungal, and viral infections. The other major problem is when a donor's stem cells (also called the graft) find that the patient's cells ( the host cells) are not the same. The donor cells may try to destroy the host's cells. The cells at high risk are those of the skin, liver and intestines. This is called graft versus host disease (GVHD) and it can be fatal.

Recently, doctors have been able to use less toxic chemotherapy treatments before patients receive their transplants. This less toxic treatment helps reduce some of the treatment related problems mentioned above. Patient's are being asked to be involved in a research study that uses this approach. One major risk of this low dose treatment is that the patient's body may reject the donor cells. This is called graft rejection. This study is designed to see if this low dose treatment is safe and effective.

This treatment plan adds CAMPATH 1H (a special protein called an antibody) to a low dose chemotherapy regimen. After chemo, the patient will receive an allogeneic (cells come from a donor) stem cell transplant. Adding CAMPATH 1H to the transplant medicines may help in treating the disease. CAMPATH 1H may reduce life-threatening and treatment related side effects like GVHD. CAMPATH 1H stays active in the body for a long time which means it may work longer to prevent GVHD. CAMPATH 1H destroys lymphocytes, a type of white cells that help fight infection, and this helps prevent graft rejection.

We want to see if the addition of CAMPATH 1H to the patient's pre-transplant low dose chemotherapy will decrease the side effects from an allogeneic stem cell transplant, while providing a curative treatment for patients with blood disorders.

DETAILED DESCRIPTION:
We expect that the patient's participation in this study will last approximately 18 months to 2 years.

Before treatment begins, they will be evaluated to confirm they meet the requirements of this study. The evaluation includes HIV testing, HIV (Human Immunodeficiency Virus) is the virus that causes Acquired Immune Deficiency Syndrome (AIDS). If the patient is HIV positive, they will not be able to be treated on this protocol.

The patient will need to have a central line. This is a thin plastic catheter or tube that is placed during surgery into one of the large veins in the chest or neck. Central lines are used to give medications IV (intravenous, by vein) or to take blood samples without having to endure frequent needle sticks.

After admission to the hospital the subject will receive:

Day -6: a single dose of total body irradiation

Day -5 to Day -2 Chemotherapy: Fludarabine plus Campath 1H through a catheter inserted into a vein (IV)

Day -2: FK506 given IV over a 24 hour period until the patient can take medication by mouth. When they can take oral medication they will take this medication by mouth every 12 hours.

Day -1 : a day of rest

Day 0: the stem cell transplant (infusion) will be given

Day +7: G-CSF will be given by subcutaneous injection until your white blood cells (granulocytes) are greater than 1000/ul.

After transplantation, they will be evaluated as follows. Routine history, physical examination, blood tests and radiology studies will be done as needed for clinical care. Bone marrow aspirate and biopsy will be done on or about day 30, 60 and 100, 180 and then yearly and as needed.

ELIGIBILITY:
INCLUSION CRITERIA:

* Myelodysplastic syndrome with IPSS score > 0.(Appendix B) Or
* Myeloproliferative disorders

  * Primary Myelofibrosis with Lile score of 1 or 2 (Appendix C)
  * Polycythemia Vera or Essential Thrombocythemia transformed to AML or Myelofibrosis and PV "spent phase" or
* Acute myelogenous leukemia or
* Chronic myelogenous leukemia
* Available Healthy Donor without any contraindications for donation. 5/6 or 6/6 related donor or 5/6 or 6/6 unrelated donor (molecular typing for DRB1)
* Able to give informed consent

EXCLUSION CRITERIA:

* Patient is pregnant or lactating or unwilling to use contraceptives.
* HIV positive patient
* Uncontrolled intercurrent infection
* Unstable angina and uncompensated congestive heart failure (Zubrod of 3 or greater)
* Severe chronic pulmonary disease requiring oxygen (Zubrod of 3 or greater)
* Hemodialysis dependent.
* Active hepatitis or cirrhosis with total bilirubin, SGOT, and SGPT greater than 3 x normal.
* Concurrent solid organ malignancy not in remission, except for Stage 0 or A prostate cancer.
* Unstable cerebral vascular disease or recent hemorrhagic stroke (less than 6 months)
* Active CNS disease from hematological disorder.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2001-12; Primary Completion 2006-09 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Day 100 Non-relapse mortality, | 100 days
  Safety and feasibility of submyeloablative conditioning as a preparative regimen for blood stem cell transplantation
Day 100 graft rejection | 100 days
  Safety and feasibility of submyeloablative conditioning as a preparative regimen for blood stem cell transplantation

SECONDARY OUTCOMES:
1 year disease free survival | 1 year
Complete Remission at 100 days | 100 days

CONTACTS AND LOCATIONS:
Overall Officials: George Carrum, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Texas Children's Hospital, Houston, Texas
  - The Methodist Hospital, Houston, Texas